CLINICAL TRIAL: NCT02790216
Title: Phase II Study of Focused Dose Painted I-125 Brachytherapy for Low to Intermediate Risk Prostate Cancer Using Deformable Registration of Multi-parametric MRI (Magnetic Resonance Imaging) to Intra-operative TRUS (Trans Rectal Ultrasound)
Brief Title: Deformable Registration of Multi-parametric MRI to Intra-operative Transrectal Ultrasound for Prostate Brachytherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-15-2845-ZS-CTIL
Record Dates: First submitted 2016-05-06; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer
Keywords: Image guided brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsies will be obtained using a transperineal approach
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brachytherapy: men eligible for monotherapy seed implant brachytherapy
  Interventions: Procedure: Brachytherapy

INTERVENTIONS:
Procedure: Brachytherapy — Biopsies will be obtained after intraoperative plan to rule out significant cancer outside a high risk planning target volume

SUMMARY:
Objective:

To focus the high dose radiation to the gross tumor in the prostate while maintaining adequate dose for control of microscopic disease elsewhere in the prostate.

In order to test the incorporation of the robust MRI and TRUS fusion algorithm in the clinical setting the investigators planned a study of Focused therapy with a primary endpoint of accurate localization of the high risk region. This is a pilot study of dose painted permanent I-125 seed implant to verify absence of tumor cells outside a high risk region using multi-parametric MRI and deformable TRUS registration. The high risk region will be dose painted to 160 Gy and the rest of the prostate will receive the normal prescription dose.

DETAILED DESCRIPTION:
Primary end-point:

Feasibility of dose painting will be determined by the absence of tumor outside the high-risk region on an intra-operative trans-perineal biopsy.

Frozen sections will not be obtained, however on receipt of the final pathology 2-4 weeks after the procedure 2 possible scenarios arise:

1. There is no evidence of cancer: this confirms the accuracy of the TRUS MRI registration.
2. There is evidence of tumor on the stereotactic biopsy: In this case a regular dosimetric check (this is performed in the Standard of care procedure and is known as post-operative dosimetry) will be performed to determine whether adequate dose was delivered. If not, as the involved needle position was recorded in the treatment plan and labeled with co-ordinates, the regular possibility of accurately adding radioactive seeds is possible.

ELIGIBILITY:
Inclusion Criteria:

* Men suitable for monotherapy with permanent Iodine 125 implant

  * Age > 50 yrs
  * PS 0-2 (WHO)
  * Histologic diagnosis of prostate adenocarcinoma made on transrectal guided prostate biopsy with no fewer than 12 cores taken
  * No more than 50% of cores involved (summary)
  * MRI of Prostate with Diffusion Weighted Imaging and Dynamic Contrast Enhancement with demonstrable lesion compatible with biopsy result
  * Gleason sum no greater than 3+4 =7 in any core
  * Clinical T stage no higher than T T (tumor) 2A
  * Prostate volume ≤60 cc
  * Serum prostate-specific antigen (PSA) no higher than 15 ng/mL
  * No prior history of malignancy except non-melanoma skin cancer
  * Must be suitable for general or spinal anesthesia

Exclusion Criteria:

Have anesthesia surgical assignment category IV or greater

* Cannot cease anti-coagulant therapy
* Had a malignancy, other than prostate or skin cancer (except malignant melanoma), within 5 years
* urethral stricture
* Prior prostate cancer therapies

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men eligible for prostate brachytherapy
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a positive biopsy outside the defined High risk Planning Target Volume | Pathological report due one month after brachytherapy implant
  Negative biopsy outside the high risk planning target volume will confirm the accuracy of the MRI TRUS elastic fusion algorithm to locate the tumor

SECONDARY OUTCOMES:
Biochemical failure as determined by Prostate specific antigen greater than nadir+2 ng/ml | 3 years
Urinary , Sexual ,Bowel and Vitality function domains | 6 months and then at years one , two and three
  Expanded Prostate Inventory Composite (EPIC)

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Symon, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Sheba_Medical_Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: Undecided